CLINICAL TRIAL: NCT06589336
Title: SUSTAIN: Promoting Sustained Behavior Change and Nutrition Security in Medicaid-Enrolled Individuals With Stage 2 Cardiovascular-Kidney-Metabolic Syndrome (CKMS)
Brief Title: SUSTAIN: Behavior Change and Nutrition Security for CKMS
Acronym: SUSTAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Joshua Joseph, MD, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023H0456
Record Dates: First submitted 2024-03-25; First posted 2024-09-19 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Stage 2 Cardiovascular-Kidney-Metabolic Syndrome; Cardiovascular Disease Other
Keywords: CKMS; Cardiometabolic Health; Cardiovascular-Kidney-Metabolic Health; Cardiovascular-Kidney-Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Other): Weeks 1-8: The intervention group will receive Instacart groceries (voucher + delivery fees), access to the Mid-Ohio Farmacy Program, behavioral nutrition counseling, and social needs screening and referrals.
  Weeks 9-16: The intervention group will receive Instacart groceries (delivery fees only), access to Mid-Ohio Farmacy program, behavioral nutrition counseling and social needs screening and referrals.
  Weeks 17-24: The intervention group will receive Instacart access (no financial support), access to the Mid-Ohio Farmacy Program and social needs screening and referrals.
  Interventions: Other: Dietary changes via Instacart vouchers; Other: Dietary changes via access to Mid-Ohio Farmacy; Other: Behavior changes via access to Health Impact Ohio Hub; Other: Behavioral nutrition counseling; Other: Cooking classes; Other: Dietary changes to Delivery fees
- Control Group (Other): Weeks 1-8: The control group will receive Instacart groceries (voucher + delivery fees) and access to the Mid-Ohio Farmacy program.
  Weeks 9-16: The control group will receive Instacart groceries (delivery fees only) and access to the Mid-Ohio Farmacy program.
  Weeks 17-24: The control group will receive Instacart access (no financial support) and access to the Mid-Ohio Farmacy program.
  Interventions: Other: Dietary changes via Instacart vouchers; Other: Dietary changes via access to Mid-Ohio Farmacy; Other: Dietary changes to Delivery fees

INTERVENTIONS:
Other: Dietary changes via Instacart vouchers — Instacart will provide consumers with the dignity of choice to shop at preferred retail stores, which is key for our behavioral change strategy. Delivery and service fees will be waived for patients, so 100% of the vouchers will be applied to groceries (all food products excluding alcohol and tobacco). The investigators will use a custom study store front with an integrated website and email option.
Other: Dietary changes via access to Mid-Ohio Farmacy — Mid-Ohio Farmacy will provide healthy food provisions through a network of food banks with fresh produce and other items.
Other: Behavior changes via access to Health Impact Ohio Hub — Health Impact Ohio Hub is a regional coordination entity that has connections with community care agencies that employ community health workers to assess social needs and make connections to resources to address social needs. The community health workers will conduct an initial needs assessment, and guide the participant through appropriate care pathways to address social needs.
  Arms: Intervention Group
Other: Behavioral nutrition counseling — All dietary recommendations will be individualized and informed by existing guidelines to improve diet quality and cardiovascular health through the Mediterranean Diet.
  Arms: Intervention Group
Other: Cooking classes — Registered dietician nutritionists will also lead cooking demonstrations every 2 weeks, focused on culinary education and building engagement among SUSTAIN participants.
  Arms: Intervention Group
Other: Dietary changes to Delivery fees — Delivery fees will be supported for SUSTAIN participants.

SUMMARY:
To determine the feasibility and engagement of participants in the SUSTAIN intervention compared to enhanced usual care over 24 weeks through mixed-methods measurement of participant enrollment, adherence, retention, and engagement (counseling, screenings, referrals, and uptake). Methods: Leveraging rigorous quantitative and qualitative evaluation, the study team will identify mechanisms driving intervention feasibility and engagement. Hypothesis: SUSTAIN will be feasible with a high degree of engagement among Medicaid-enrolled participants with Stage 2 CKMS in comparison to enhanced usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be Medicaid enrolled, and/or dual enrolled in Medicaid
* Patients must be diagnosed with at least one of the following diseases: hypertension, type 2 diabetes mellitus, hyperlipidemia, chronic kidney disease and/or metabolic syndrome
* Patients must at least 18 years of age or older at the time of signing consent
* Patient must have access to internet-enabled device
* Patient has no objections to online grocery shopping, home food deliveries, or nutrition counseling
* Patient lives in setting able to receive Instacart deliveries (e.g., non-institutionalized)
* Patient is willing to use a credit card for Instacart back-up payments

Exclusion Criteria:

* Have any condition that impacts digestion, metabolism, or food intake (e.g., surgical loss of esophagus, stomach, or colon, pancreatic dysfunction, bariatric surgery, brain surgery that alters cognition, etc.)
* Have active digestive illnesses (i.e., Celiac disease, irritable bowel syndrome, chronic malabsorption)
* Any comorbidity such as psychiatric or general illness that may put the subject at risk as determined by investigator
* Any other factor which, in the investigator's opinion, is likely to compromise the subject's ability to participate in the study
* Recent (e.g., 6 months) participation in other behavioral nutrition trials
* Are currently pregnant or are planning to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Enrollment | Week 1
  Enrollment will be determined by the percent of eligible participants who enroll in the study.
Adherence - Mid-Ohio Farmacy | 24 weeks
  Adherence will be determined based on the number of visits to food pantries divided by the total number of possible visits.
Adherence - Health Impact Ohio | 24 weeks
  Adherence to the Health Impact Ohio component of the intervention to address social needs will be determined based on the percent of participants that enroll with the community health worker.
Adherence - Behavioral Nutritional Counseling | 16 weeks
  Adherence to behavioral nutritional counseling will be determined by the number of interactions with behavioral counseling out of the total number of counseling sessions offered.
Retention | 24 weeks
  The percent of participants that complete the study visits at 12 and 24 weeks.
Engagement | 8 weeks
  Engagement will be determined by the amount of total dollars spent on Instacart per participant.

SECONDARY OUTCOMES:
Nutrition Security | 24 weeks
  Nutrition security will be measured using the Center for Nutrition and Health Impact Nutrition Security Screener. The screener has 4 questions with score ranging from Never = 4, Rarely = 3 Sometimes = 2, Often = 1, Always = 0. The 4 question scores are averaged for a final score. Higher scores indicate a greater degree of Household Nutrition Security.
Dietary Patterns | 24 weeks
  Mediterranean Eating Pattern for Americans (MEPA) Version III will be used to assess changes in the MEPA. The MEPA screener includes 21 questions on the consumption of foods typical of the Mediterranean diet as well as fast food, convenience foods, and sugar-sweetened beverages. The total MEPA-III score ranges from 0 to 21 (higher scores indicate greater intakes of Mediterranean foods). Change in MEPA Scores at 24-week follow-up will be calculated using between-subject differences, using a linear mixed-effects to evaluate changes from baseline in MEPA score (range 0-21, higher scores are better).
Cardiometabolic Health | 24 weeks
  American Heart Association Life Essential 8 will be calculated with a range of 0-100 to measure cardiometabolic health. Change in cardiometabolic health at 24-week follow-up will be calculated using between-subject differences, using a linear mixed-effects to evaluate changes from baseline in Life's Essential 8 score (range 0-100, higher scores are better).
Purchasing Behavior | 24 weeks
  Purchasing behavior will be analyzed by measuring the types of food purchased using receipts from instacart. The instacart receipts will be coded into categories of food consistent with a Mediterranean healthy eating pattern (i.e. fruits, vegetables, nuts, etc.) and changes will be evaluated over the 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Joseph, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No